CLINICAL TRIAL: NCT05671861
Title: Design of a Low-Cost Therapeutic Device for Patients With Radiation-Related Trismus
Brief Title: Evaluating a Low-Cost Therapeutic Device in Managing Head and Neck Cancer Patients With Radiation-Related Trismus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mount Zion Health Fund (Other); American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22206; NCI-2022-10268 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Trismus; Head and Neck Cancer
Keywords: Radiation-related
MeSH Terms: conditions — Trismus; Head and Neck Neoplasms | interventions — Equipment and Supplies; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Part I (medical device usage, questionnaire) (Experimental): Each participant will complete a single 45-minute visit in which consists of questionnaires about features that are important to them in trismus treatment, test a prototype of a trismus therapy device, and complete an online feedback questionnaire about their experience using the device.
  Interventions: Device: Trismus Device Prototype; Other: Questionnaires
- Part II (medical device usage, mobile app usage) (Experimental): Participants will be asked to use the device at least three times per week and up to daily for a period of 15-20 minutes over 6 weeks. Participants will be evaluated at baseline, at the 3-week (halfway) visit, and at the end of the 6-week treatment period under supervision of a speech language pathologist on study. Participants will then utilize a mobile app to help track treatment progress.
  Interventions: Device: Trismus Device Prototype; Other: Mobile Application

INTERVENTIONS:
Device: Trismus Device Prototype — Device is noninvasive and will be inserted between patient's upper and lower teeth
  Other Names: Medical Device
Other: Questionnaires — Surveys will be administered to participants
  Other Names: Survey Administration
  Arms: Part I (medical device usage, questionnaire)
Other: Mobile Application — A study-specific, accompanying secure mobile application for users to track progress will be created.
  Other Names: Mobile App
  Arms: Part II (medical device usage, mobile app usage)

SUMMARY:
This trial evaluates how well a new therapeutic device works in managing trismus in patients who received radiation treatment for head and neck cancer. Radiation therapy is a common form of treatment in patients with head and neck cancers. However, changes to surrounding tissue following radiation therapy may lead to trismus, an inability to open the mouth fully. This can create significant functional impairment leading to malnutrition due to impaired chewing, risk of dental infections due to impaired oral hygiene, difficulty with speech, and decreased health-related quality of life. Exercise therapy is the mainstay of treatment for post-radiation trismus to help improve mobility and flexibility and increase range of mouth opening. This new device is non-invasive and is similar to other jaw stretching devices where a mouthpiece is placed between the teeth and a hand-lever is used to spread open the upper and lower jaw. However, it will also have additional sensors to measure pressure exerted by the hands and jaw as well as the distance to open the mouth which could help guide therapy. This study may help doctors customize a device to patient-specific needs, provide real-time feedback, and encourage compliance for trismus exercise therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the clinical efficacy of the trismus device, as measured by the change in maximum interincisal opening over the six-week treatment period.

SECONDARY OBJECTIVE:

I. To assess participants compliance rates and jaw opening pressures when using this device.

OUTLINE: Participants are assigned to 1 of 2 parts.

PART I: Participants test the trismus device and complete questionnaires on study.

PART II: Participants undergo exercise therapy with the trismus device under supervision of a speech language pathologist on study.

Participants will be on study for up to 6 weeks with a follow-up visit 7 days after completion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age at visit 1.
* Documentation of a radiation-induced trismus diagnosis as evidenced by one or more clinical features consistent with the trismus phenotype (maximum interincisal opening (MIO) < 35 mm) and a history of head and neck radiation
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.
* Minors (age < 18 years) or patients with inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in maximum interincisal opening (MIO) over time | Up to 6 weeks
  The mean change in MIO from baseline to end of treatment at 6 weeks will be reported

SECONDARY OUTCOMES:
Number of participants with device-related adverse events | Up to 1 year
  During the study, research staff consisting of trained speech language pathologists will monitor patients undergoing exercise therapy for any adverse events. Adverse events for the eligible population will include the number of patients for whom the event occurred by the severity and relationship to study device. Adverse event rates will be coded by body system and Medical Dictionary for Regulatory Activities (MedDRA) classification term and graded using the CTCAE grading scale of (1) Mild to (5) Death.
Rate of compliance | Up to 1 year
  Percentage of participants who utilize the addition of the study-specific mobile application designed to track participant progress and participant compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Park, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No